CLINICAL TRIAL: NCT05398679
Title: Oral Antimicrobial Treatment vs. Outpatient Parenteral for Infective Endocarditis
Acronym: OraPAT-IEGAMES
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fundacion Clinic per a la Recerca Biomédica (Other)
Responsible Party: Principal Investigator, Anna Cruceta, Project Manager Clinical Trial Unit, Fundacion Clinic per a la Recerca Biomédica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OraPAT-IE GAMES
Record Dates: First submitted 2022-05-04; First posted 2022-06-01 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Endocarditis Infective
MeSH Terms: conditions — Endocarditis | interventions — Cefaclor; Ciprofloxacin; Clindamycin; Dicloxacillin; Dosage Forms; Injections; Levofloxacin; Linezolid; Moxifloxacin; Sulfamethoxazole; Trimethoprim; Trimethoprim, Sulfamethoxazole Drug Combination; tedizolid; Amoxicillin

STUDY DESIGN:
Intervention Model Description: National multi-center study, open, controlled, and randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OPAT (Active Comparator): Patients with infective endocarditis diagnostic, who have completed at least 10 days of intravenous therapy, and/ or seven days in the case of cardiac valvular surgery, and shown good clinical evolution and no clinical or echocardiographic signs of potential bad prognosis will be randomized. If assigned to this arm the patient will recieve parenteral antibiotics until the end of treatment.
  Interventions: Drug: Cefaclor; Drug: Ciprofloxacin Injection; Drug: Clindamycin Injection; Drug: Dicloxacillin; Drug: Fusidic Acid Only Product in Parenteral Dose Form; Drug: Levofloxacin Injection; Drug: Linezolid Injectable Product; Drug: Moxifloxacin Injectable Product; Drug: Rifampicin Only Product in Parenteral Dose Form; Drug: Sulfamethoxazole / Trimethoprim Injectable Product; Drug: Tedizolid Injection; Drug: Amoxicillin
- Oral Therapy (Experimental): Patients with infective endocarditis diagnostic, who have completed at least 10 days of intravenous therapy, and/ or seven days in the case of cardiac valvular surgery, and shown good clinical evolution and no clinical or echocardiographic signs of potential bad prognosis will be randomized. If assigned to this arm the patient will recieve oral antibiotics until the end of treatment.
  Interventions: Drug: Ciprofloxacin Tablets; Drug: Clindamycin Oral Capsule; Drug: Dicloxacillin Oral Capsule; Drug: Fusidic Acid Only Product in Oral Dose Form; Drug: Levofloxacin Oral Tablet; Drug: Linezolid Oral Tablet; Drug: Moxifloxacin tablet; Drug: Rifampicin Only Product in Oral Dose Form; Drug: Sulfamethoxazole / Trimethoprim Oral Tablet [Bactrim]; Drug: Tedizolid Oral Tablet; Drug: Amoxicillin Capsules; Drug: Cefaclor Capsules

INTERVENTIONS:
Drug: Cefaclor — cefaclor intravenous 2 gr/day
  Arms: OPAT
Drug: Ciprofloxacin Tablets — 500-750 mg/12 hrs (maximum 3g x day)
  Arms: Oral Therapy
Drug: Ciprofloxacin Injection — 1200 mg/day maximum dose IV
  Arms: OPAT
Drug: Clindamycin Oral Capsule — 600 mg/8 hours (maximum 1.800 mg x day)
  Arms: Oral Therapy
Drug: Clindamycin Injection — 600 mg/8 hours (maximum 1.800 mg x day) IV
  Arms: OPAT
Drug: Dicloxacillin Oral Capsule — 1g/8 hours (maximum 4 gr day)
  Arms: Oral Therapy
Drug: Dicloxacillin — 1g/8 hours (maximum 4 g x day) IV
  Arms: OPAT
Drug: Fusidic Acid Only Product in Oral Dose Form — 0,750g/12 hours (maximum 1,5 g x day)
  Arms: Oral Therapy
Drug: Fusidic Acid Only Product in Parenteral Dose Form — 0,75 g/12 hours (maximum 1,5 g x day)
  Arms: OPAT
Drug: Levofloxacin Oral Tablet — 0.5g/12-24hours (maximum 1 g x day)
  Arms: Oral Therapy
Drug: Levofloxacin Injection — 0.5g/12-24hours (maximum 1 g x day)
  Arms: OPAT
Drug: Linezolid Oral Tablet — 0,6 g/12 hours (maximum 1200 mg x day)
  Arms: Oral Therapy
Drug: Linezolid Injectable Product — 0,6 g/12 hours (maximum 1200 mg x day)
  Arms: OPAT
Drug: Moxifloxacin tablet — 0,4 g/day (maximum 400 mg x day)
  Arms: Oral Therapy
Drug: Moxifloxacin Injectable Product — 0,4 g/day (maximum 400 mg x day)
  Arms: OPAT
Drug: Rifampicin Only Product in Oral Dose Form — 0,3-0,5 g/12 hours (maximum 1200 mg x day)
  Arms: Oral Therapy
Drug: Rifampicin Only Product in Parenteral Dose Form — 0,3-0,6 g/12 hours (maximum 1200 mg x day)
  Arms: OPAT
Drug: Sulfamethoxazole / Trimethoprim Oral Tablet [Bactrim] — sulfamethoxazole 1600 mg/trimethoprin 320 mg (maximum x day)
  Arms: Oral Therapy
Drug: Sulfamethoxazole / Trimethoprim Injectable Product — sulfamethoxazole 1600 mg/trimethoprin 320 mg (maximum x day)
  Arms: OPAT
Drug: Tedizolid Oral Tablet — 200 mg tedizolid (maximum x day)
  Arms: Oral Therapy
Drug: Tedizolid Injection — 200 mg (maximum x day)
  Arms: OPAT
Drug: Amoxicillin Capsules — 1 gr/6 hours (4 g x day)
  Arms: Oral Therapy
Drug: Amoxicillin — 1 gr/6 hours (4 g x day) Intravenous
  Arms: OPAT
Drug: Cefaclor Capsules — 2 gr/day
  Arms: Oral Therapy

SUMMARY:
Non-inferiority trial to determine whether partial oral treatment is non-inferior to OPAT(Outpatient parenteral therapy) in patients diagnosed with infective endocarditis

DETAILED DESCRIPTION:
The trial will include patients diagnosed with left-side Infective Endocarditis according to the modified Duke criteria, with ≥10 days of appropriate parenteral antibiotic treatment overall and at least one week of appropriate parenteral treatment after valve surgery

The patients will be randomized in two arms, one with oral antibiotic therapy and the other one with outpatient parenteral therapy

This trial aims to demonstrate the non-inferiority of outpatient oral antibiotic therapy in comparison with outpatient parenteral antibiotic treatment (OPAT), to improve the quality of life of infective endocarditis (IE) patients, and to reduce the cost of the intervention without increasing morbidity and mortality rates

ELIGIBILITY:
Inclusion Criteria:

* Left-sided native or prosthetic infective endocarditis based on the modified Duke criteria infected with one of the following nonresistant microorganisms: Non-resistant streptococci and other gram positive cocci,e.g., Granulicatella and Abiotrophia; Enterococcus faecalis; Staphylococcus aureus;coagulase-negative staphylococci and HACEK group.
* Male or female 18 years old or older.
* 10 days or more of appropriate parenteral antibiotic treatment overall and at least one week of appropriate parenteral treatment after value surgery.
* Temperature inferior to 38ºC for more than two days. 5. C-reactive protein dropped to <25% of peak value or <20 mg/l, and white blood cell count <15x10^9/l during antibiotic treatment
* Transthoracic / transesophageal echocardiography performed within 48 hours of randomization

Exclusion Criteria:

* Body mass index >40
* Concomitant infection requiring intravenous antibiotic therapy
* Inability to give informed consent to participation
* Suspicion of reduced absorption of oral treatment due to abdominal disorder
* Microorganisms with no oral combinations for treatment (two active antibiotics of different families)
* Any immunosuppressive disease or any medical condition at the discretion of the investigator that may preclude oral or OPAT therapy
* No family or appropriate home support
* Reduced compliance
* Women of childbearing potential with a positive pregnancy test, or participants (male or female) who wish to plan a pregnancy during the trial period
* Women in lactancy period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-08-17 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
Non-inferiority of outpatient oral vs parenteral antibiotic therapy measured by the number of unplanned hospitalizations | At any time during the study duration (up to 24 months)
Non-inferiority of outpatient oral vs parenteral antibiotic therapy measured by the number of all-cause mortality | At any time during the study duration (up to 24 months)
Non-inferiority of outpatient oral vs parenteral antibiotic therapy measured by the number of relapses of Infective Endocarditis | within 6 months from diagnosis of Infective Endocarditis
Non-inferiority of outpatient oral vs parenteral antibiotic therapy measured by the number of patients requiring cardiac surgery | At any time during the study duration (up to 24 months)

SECONDARY OUTCOMES:
Quality of life and patient satisfaction of infective endocarditis patients. It will be measured through the standardized Saillen questionnaire of antibiotic treatment satisfaction | At any time during the study duration (up to 24 months)
Costs of both interventions, measured through a pharmaco-economic sub-study including direct and indirect costs, following the methodology described by Lacroix A et al Med Mal Infect. 2014 | At any time during the study duration (up to 24 months)
  through a pharmacoeconomic analysis
The complications related to parenteral and oral administration of antibiotics will be measured through the number of antibiotic adverse reactions, catheter-related adverse events, and number of superinfections | At any time during the study duration (up to 24 months)
  such as antibiotic or catheter-related adverse events e.g.,phlebitis and line-related bloodstream infections, and superinfections

CONTACTS AND LOCATIONS:
Locations (20):
- Spain (20):
  - Hospital Virgen de la Macarena, Seville, Andalusia
  - Hospital Virgen del Rocío, Seville, Andalusia
  - Hospital Son Espases, Palma de Mallorca, Balearic Islands
  - Parc Taulí Hospital Universitari, Sabadell, Barcelona
  - Hospital Mútua de Terrassa, Terrassa, Barcelona
  - Hospital Universitario de Cruces, Barakaldo, Bizcaia
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital Universitario de Donostia, Donostia / San Sebastian, Guipuzcoa
  - Hospital San Pedro, Logroño, La Rioja
  - Hospital Virgen de Arrixaca, El Palmar, Murcia
  - Hospital universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital General de Alicante, Alicante
  - Hospital del Mar, Barcelona
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Sant Pau, Barcelona
  - Hospital Bellvitge, Barcelona
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Ramón y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitari i Politècnic La Fe, Valencia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Cuervo G, Hernandez-Meneses M, de Alarcon A, Luque-Marquez R, Alonso-Socas MM, Lopez-Lirola A, Gonzalez-Ramallo V, Goikoetxea-Agirre AJ, Nicolas D, Goenaga MA, Merino E, Escrihuela-Vidal F, Martin-Davila P, Loeches B, Boix-Palop L, Gasch O, Camprecios M, Hernandez-Torres A, Garcia-Alvarez L, Pajaron M, Ribas MA, Blanes-Hernandez R, Lopez-Montesinos I, Lopez-Cortes LE, Vidal B, Fernandez-Pittol M, Navarro D, Moreno A, Sala C, Ambrosioni J, Miro JM; OraPAT-IE GAMES Investigators. Oral vs. Outpatient Parenteral Antimicrobial Treatment for Infective Endocarditis: Study Protocol for the Spanish OraPAT-IE GAMES Trial. Infect Dis Ther. 2025 Mar;14(3):643-655. doi: 10.1007/s40121-025-01110-9. Epub 2025 Mar 1. PMID 40024946